CLINICAL TRIAL: NCT07304102
Title: Assessment of GORE® EXCLUDER® IBE Plus Stent Graft Performance in Patients Undergoing Endovascular Iliac Revascularization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBE 25-05
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Common Iliac Artery Aneurysm; Aorto Iliac Aneurysm
Keywords: EVAR Revision; EVAR; Endovascular Aneurysm Repair; AIAA; CIAA; IBE; Iliac Aneurysm
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Arm (Experimental): Subjects representative of AIAA/ CIAA pathology to be treated with IBE Plus Stent Graft
  Interventions: Device: GORE® EXCLUDER® IBE Plus Stent Graft
- Secondary Arm (Experimental): Subjects representative of EVAR revision to be treated with IBE Plus Stent Graft
  Interventions: Device: GORE® EXCLUDER® IBE Plus Stent Graft

INTERVENTIONS:
Device: GORE® EXCLUDER® IBE Plus Stent Graft — Endovascular aneurysm repair with the GORE® EXCLUDER® IBE Plus Stent Graft

SUMMARY:
The IBE 25-05 study will be a prospective, non-randomized, multicenter, interventional two arm evaluation designed to assess the safety and effectiveness of the GORE® EXCLUDER® IBE Plus Stent Graft in patients with common iliac artery aneurysm (CIAA) or aorto-iliac aneurysm (AIAA) disease.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the safety and effectiveness of the GORE® EXCLUDER® IBE Plus Stent Graft for endovascular revascularization in patients with common iliac artery aneurysm (CIAA) or aorto-iliac aneurysm (AIAA) disease requiring intervention. The study population includes adults aged 22 years and older, both male and infertile female, who meet specific anatomical criteria.

The main questions it aims to answer are:

Does the IBE Plus Stent Graft provide clinical benefit and maintain safety? Does the device maintain effectiveness?

Researchers will evaluate two parallel study arms:

* Primary Arm: Subjects with AIAA/CIAA pathology, including a subset newly eligible for treatment with IBE Plus.
* Secondary Arm: Subjects requiring EVAR revision for previously treated AIAA/CIAA.

Participants will:

* Undergo pre-procedure assessments (informed consent, physical exam, lab tests, and CTA imaging).
* Receive endovascular treatment with the IBE Plus Stent Graft.
* Attend follow-up visits at 1, 6, 12, 24, 36, 48, and 60 months post-procedure for physical exams, lab tests, and imaging.
* Be monitored for adverse events, device performance, and need for reintervention.

ELIGIBILITY:
Primary Arm Inclusion Criteria

The subject is / has:

1. The target lesion and surrounding vasculature are amenable to treatment with IBE Plus system requirements:

   1.1. Common iliac artery to be treated must have a common iliac diameter ≥ 25 mm with or without concomitant abdominal aortic aneurysm 1.2. Minimum diameter ≥ 12 mm within the proximal implantation zone of IBE Plus as assessed by flow lumen; calcium excluded 1.3. Intended treatment length must be ≥ 100 mm in unilateral application or a combination of ≥ 100 mm and ≥ 150 mm in bilateral application 1.4. The planned distal target landing zone within the internal iliac artery is within the trunk of the internal iliac artery with at least 15 mm of seal zone 1.5. Iliac vasculature meets anatomical specifications for selected VBX Stent Graft(s)
2. Aortoiliac vasculature meets anatomical specifications for selected EXC or EXCC Devices
3. Informed Consent Form (ICF) is signed by subject
4. Subject is capable of complying with protocol requirements, including follow-up
5. Life expectancy > 2 years
6. Age ≥ 22 years at time of informed consent signature
7. Male or infertile female

Secondary Arm Inclusion Criteria

The subject is / has:

1. Present with any one of the following treatment indications:

   1.1. The subject has a confirmed Type Ib endoleak of a previously implanted Gore EVAR device where its distal portion within the common iliac artery has a luminal diameter of at least 12 mm. Minimum diameter of ≥ 12 mm within the proximal implantation zone of IBE Plus as assessed by flow lumen; calcium excluded 1.2. The subject has documented diameter growth of the common iliac artery of at least ≥ 5 mm in the presence of a previously implanted Gore EVAR device where its distal portion within the common iliac artery has a luminal diameter of at least 12 mm. The planned distal target landing zone within the internal iliac artery is within the trunk of the internal iliac artery with at least 15 mm of seal zone
2. Aortoiliac vasculature meets anatomical specifications for selected EXC or EXCC Devices
3. Informed Consent Form (ICF) is signed by subject
4. Subject is capable of complying with protocol requirements, including follow-up
5. Life expectancy > 2 years
6. Age ≥ 22 years at time of informed consent signature
7. Male or infertile female

Primary Arm and Secondary Arm Exclusion Criteria

The subject is / has:

1. Mycotic or ruptured aneurysm
2. ASA class V (moribund patient not expected to live 24 hours with or without operation)
3. Renal insufficiency defined as creatinine > 1.8 mg/dL or undergoing dialysis
4. NYHA class IV
5. Dissected, heavily calcified, or heavily thrombosed landing zone(s)
6. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
7. Participating in another investigational drug or medical device study within one year of study enrollment
8. An active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication) that may place the patient at increased risk of endovascular infection. Subjects with a chronic infection (such as HIV, Hepatitis C, etc.) that is well controlled under their current treatment regimen may be eligible
9. Degenerative connective tissue disease, e.g., Marfan's or Ehler-Danlos Syndrome
10. Planned concomitant surgical procedure or major surgery within 30 days of treatment date
11. History of drug abuse, e.g., cocaine or amphetamine, within 1 year of treatment
12. Known sensitivities or allergies to the device materials

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Freedom From Composite of the Following: All-Cause Mortality, Serious Stroke, Myocardial Infarction, Bowel Ischemia, Paraplegia, Respiratory Failure, Renal Function Decline, Conversion to Open Surgical Repair | Through 30 days post-treatment
  Freedom from composite of any of the following events:
  * All-cause mortality
  * Serious stroke
  * Myocardial infarction
  * Bowel ischemia requiring surgical resection or not resolving with medical therapy
  * Paraplegia (grade 3)
  * Respiratory failure requiring prolonged (>24 hours from anticipated) mechanical ventilation or reintubation
  * Renal function decline resulting in >50% reduction in baseline eGFR or new-onset dialysis
  * Conversion to open surgical repair
Freedom From Composite of the Following: IBE Plus-Related Reinterventions Involving Type Ib / Ic or Type III Endoleak, Total Occlusion of Any IBE Plus Component, Loss of Primary Patency of the Internal Iliac Device Component | Through the 6 month follow-up visit
  Composite of the following events:
  * IBE Plus-related reinterventions involving Type Ib / Ic or Type III endoleak
  * Total occlusion of any IBE Plus component
  * Loss of primary patency of the internal iliac device component

SECONDARY OUTCOMES:
Freedom From New Onset Buttock Claudication on an IBE Plus-Treated Side | Through the 6 month follow-up visit
  Freedom from new onset buttock claudication on an IBE Plus-treated side

IPD SHARING:
Plan to Share IPD: No